CLINICAL TRIAL: NCT07314892
Title: Prospective Assessment of the Impact of Psychiatric Status on Clinical Symptom Severity in Patients With Graft-versus-Host Disease (GvHD).
Brief Title: Psychiatric Status and Symptom Severity in Graft-versus-Host Disease (GvHD).
Acronym: Psych-GvHD
Status: Recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Jan Puchowski, MD, Medical University of Gdansk
Other Study IDs: KB/90/2025
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: GVHD, Chronic; GVHD - Graft-Versus-Host Disease; GVHD; Quality of Life; Depression Disorders; Cognitive Impairments
Keywords: GvHD; depression; quality of life; Cognitive impairment
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease; Cognitive Dysfunction; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cGvHD and depression: Patients with chronic graft-versus-host disease (GvHD) diagnosed with depressive disorders, adjustment disorders, or cognitive impairment, diagnosed according to ICD-10 and/or DSM-5 criteria.
- cGvHD without depression: Patients with chronic graft-versus-host disease (GvHD) without a diagnosis of depressive disorders, adjustment disorders, or cognitive impairment (control group).

SUMMARY:
This prospective observational study evaluates the association between psychiatric status, GvHD-related symptom severity, and health-related quality of life in patients with graft-versus-host disease. Standardized and validated assessment tools, including the Lee Symptom Scale, will be used to collect psychiatric, clinical, and demographic data.

DETAILED DESCRIPTION:
Graft-versus-host disease (GvHD) is a significant complication following allogeneic hematopoietic stem cell transplantation and is associated with substantial symptom burden, impaired quality of life, and increased psychiatric morbidity. Despite its clinical relevance, the relationship between psychiatric status and the severity of GvHD-related symptoms remains insufficiently characterized.

This prospective observational study aims to systematically assess psychiatric status, symptom severity, and health-related quality of life in patients with GvHD using standardized and validated instruments. Demographic and clinical data will be collected to establish a comprehensive patient registry. The study will evaluate the association between psychiatric disorders and the intensity of GvHD-related symptoms, as measured by the Lee Symptom Scale, and will explore the bidirectional relationship between depressive symptoms and the clinical course of GvHD. The findings are expected to inform the development of evidence-based recommendations for therapeutic support aimed at improving clinical outcomes and quality of life in patients with GvHD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a clinically established diagnosis of graft-versus-host disease (GvHD) receiving specialist follow-up care at the Bone Marrow Transplantation Outpatient Clinic, University Clinical Center (UCK), Gdańsk.

Exclusion Criteria:

* Severe psychiatric disorders precluding adequate cooperation, terminal-stage multiorgan failure, or refusal to provide informed consent for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 75 years, including both female and male participants, with a clinically confirmed diagnosis of graft-versus-host disease (GvHD). Participants are receiving specialist follow-up care at a bone marrow transplantation outpatient clinic and meet the predefined inclusion and exclusion criteria regarding clinical and psychiatric status.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Identification of depression as a factor associated with increased GvHD-related symptom burden and reduced health-related quality of life. | Baseline and follow-up assessments during the study period (up to 12 months).
Assessment of therapeutic benefits associated with combined antidepressant treatment and psychotherapy, antidepressant treatment alone, and psychotherapy alone. | Baseline and follow-up assessments during the study period (up to 12 months).
Support for the integration of systematic psychiatric assessment into standard multidisciplinary care protocols for patients with graft-versus-host disease. | Baseline and follow-up assessments during the study period (up to 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Puchowski, MD, Principal Investigator — Department of Hematology and Transplantology, Faculty of Medicine, Medical University of Gdańsk, Gdańsk, Poland Department of Psychiatry, Faculty of Medicine, Medical University of Gdańsk, Gdańsk, Poland; Agnieszka Piekarska, MD PhD, Principal Investigator — Department of Hematology and Transplantology, Faculty of Medicine, Medical University of Gdańsk, Gdańsk, Poland; Karol Grabowski, MD PhD, Study Director — Department of Psychiatry, Faculty of Medicine, Medical University of Gdańsk, Gdańsk, Poland
Locations (1):
- Department of Hematology and Transplantology, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No